CLINICAL TRIAL: NCT02965144
Title: Long-term Survivors of High-grade Glioma
Brief Title: Long Term Survivors of High-grade Glioma and Their Caregivers
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Karin Piil, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: LTS01
Record Dates: First submitted 2016-11-09; First posted 2016-11-16 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Quality of Life; Brain Diseases; Depression; Physical Impairment
Keywords: long-term survivors, high-grade glioma
MeSH Terms: conditions — Brain Diseases; Depression; Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HGG patients: single-group study- long term survivors
  Interventions: Other: no treatment

INTERVENTIONS:
Other: no treatment — no treatment

SUMMARY:
This study builds on the limited body of existing literature combined with the results from the investigators' previous research conducted with 30 newly diagnosed patients with high-grade glioma (HGG) and 33 of their caregivers. This research established an overview of the daily life experiences when diagnosed with a HGG or being a caregiver. Descriptions of needs and preferences from time of diagnosis to one year exist. However, such data are still lacking the representation from long-term survivors (LTS) and their caregivers.

This mixed methods study aims to address perspectives on daily life experiences of long-term survivors with HGG and their caregivers as well as the needs and preferences for support, rehabilitation and palliation.

Separate telephone interviews with patients and their caregivers and self-reported questionnaires for patients will be conducted. The mixed methods design is a convergent sequential design using an identical sampling.

DETAILED DESCRIPTION:
The dominant status relies on the qualitative data as the interviews are emphasized as the best suited method to address the primary aim of this study. The interviews follow a semi-structured interview guide for patients and for caregivers.

Information about socio-economic conditions, disease and treatment variables will be obtained by the investigator at baseline. Disease, treatment and clinical variables will be collected including the World Health Organization (WHO) performance scale (PS) which will be obtained by medical chart review. The self-reported questionnaires (quantitative data) are viewed as a useful supplemental data source, and embrace the topics as distress, anxiety and depressive symptoms.

Theoretical Framework The qualitative and quantitative research components represent different paradigmatic traditions including diverse ontological, epistemological and methodological assumptions. However, these paradigms are not necessarily incompatible. This study applied a pragmatic paradigm, reflecting a pluralistic view using both inductive and deductive reasoning. Applying a qualitative perspective, the present interviews seek to capture the subjective experiences of the study participants related to their life situation.

Analysis The semi-structured interviews will be recorded and transcribed in full length by the interviewer. Interview data will be transferred to NVivo 10 (qualitative data analysis computer software package) software program. A thematic analysis will be conducted for the analysis of the semi-structured interviews. Thematic analysis is a basic method for qualitative analysis as it identifies, analyzes and reports themes and patterns within data. The findings will be presented in themes and subthemes. A theme is an expression or context being defined as important by the researchers. In this study a theme is not necessarily dependent on quantifiable measures, but rather captures an important meaning in relation to the research questions and aims. Data from the interviews are descriptive in nature and reflect the subjective experience of the life situation of patients with HGG and their caregivers. The steps for thematic analysis are inspired by Braun and Clarke and as follows; Step 1) Data are transcribed immediately after an interview by the investigator or a research assistant. Transcriptions are read several times until the investigators are familiar with the depth and extent of the content. This process guides the investigators to the next level of analysis. Step 2) The text is read and divided into units of meanings, which are identified by the investigators. Some meaning units are sentences, others a whole paragraph. In this process data are coded in order to organize them into meaningful groups. This process assures that the whole dataset is systematically worked through by the investigators. Step 3) Then, the codes are analyzed in order to consider if different codes can be combined into mutual themes. This three step process will result in a collection of themes and sub-themes.

Statistical analysis The PS, the The Hospital Anxiety and Depression Scale (HADS) sub-scales, the The Functional Assessment of Cancer Therapy, General and brain cancer (FACT-G and FACT-Br) sub-scales and the responses to the ordinal items of the leisure time physical activity scale will be analysed separately. Socio-economic information and data from questionnaires will be entered into a database. The questionnaires will be analyzed according to their manuals. Categorical variables will be reported as frequencies and percentages, while continuous variables are reported as mean and standard deviations (s.d.) using a significance level of p\0.05. HADS and FACT-Br data refer to the normative values. The statistical analysis will be performed with SAS (Statistical Analysis System) statistical software, version 9.3.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥18 years of age, with the ability to speak and understand Danish. Caregivers are eligible if they are named by the patient as being one of the closest relative(s) providing care at home on a regular basis.

Exclusion Criteria:

* not able to speak and understand Danish
* not able to participate in being interviewed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with HGG for a minimum of 3 years and their caregivers
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Piil, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- University hospital of Copenhagen, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
The results from the thematic analysis of the interviews will be discussed with other researchers

REFERENCES:
- [Derived] Piil K, Christensen IJ, Grunnet K, Poulsen HS. Health-related quality of life and caregiver perspectives in glioblastoma survivors: a mixed-methods study. BMJ Support Palliat Care. 2022 Dec;12(e6):e846-e854. doi: 10.1136/bmjspcare-2019-001777. Epub 2019 Jun 28. PMID 31253732

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A database comprised 18 patients, who were screened; 1 declined participation due to lack of motivation and 4 were lost to follow-up during screening. A total of 13 pt were enrolled, started the study and completed the study.
Period: Overall Study
Arm/Group | HGG Patients
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: HGG patients diagnosed for more than 3 years ago
Arm/Group | HGG Patients
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years]
  Age | 56 [31 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Identifying With the Three Main Themes Identified
Description: Interviews seek to explore the perspectives on the life situation and quality of life Analysis of the interviews identified three main themes, shared by all the patients : (1) Searching for meaningful activities. (2) Selecting information that enhances self-management strategies. (3) Protection for safety reasons.
Time Frame: up to 5 months
Population: The dataset was analysed according to the steps described by Braun and Clarke in "Using Thematic analysis in psychology".
Measure: Count of Participants; unit: Participants
Groups:
- HGG Patients: single-group study- long term survivors
  no treatment: no treatment Analysis of the interviews identified three main themes, shared by patients and their caregivers: (1) Searching for meaningful activities. (2) Selecting information that enhances self-management strategies. (3) Protection for safety reasons.
Arm/Group | HGG Patients
Number analyzed (Participants) | 13
Participants | 13

2. Secondary Outcome: The Hospital Anxiety and Depression Scale (HADS)
Description: The questionnaire is divided into two sub-scales for anxiety and depression with seven questions each all; 14 questions are rated on a four-point scale representing the degree of distress [0 = none, 4 = unbearable]. The responses from HADS are presented as mean scores for anxiety and depression.
  Higher scores indicating worse outcome for depression (range 0.00-16.00) and anxiety (range 0.00-16.00).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HGG Patients
Number analyzed (Participants) | 13
units on a scale
  anxiety | 5.50 (5.17)
  depression | 4.15 (4.00)

3. Secondary Outcome: The WHO Performance Scale
Description: The Performance Scale covers a rating from 0 to 5; 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2=Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3=Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4=Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair; 5= Dead
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | HGG Patients
Number analyzed (Participants) | 13
Participants
  PS value 0 | 5
  PS value 1 | 6
  PS value 2 | 1
  PS value 3 | 1

4. Secondary Outcome: The Functional Assessment of Cancer Therapy, General (FACT-G)
Description: FACT-Br total score range 84.00-195.67 The FACT-G total score provides a summary of the overall HRQOL [range 0-108]. The higher the score, the better HRQOL.
Time Frame: Baseline
Population: Quality of life
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HGG Patients
Number analyzed (Participants) | 10
units on a scale
  FACT-G | 86.45 (20.03)
  FACT-Br | 147.71 (40.3)

5. Secondary Outcome: Questionnaire on Leisure Time Physical Activity Level
Description: 0=fully active; 1=restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2=ambulatory and capable of all self-care but unable to carry but any work activities, up and about more than 50% of waking hours; 3=capable of only limited self-care, 4=bedbound, completely disabled
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- HGG Patients: single-group study- long term survivors
  no treatment: no treatment
  Concerning depression, HADS showed moderate depressive symptoms in one patient (10%), and none of the patients reported having severe symptoms. Our data seem to be lower for anxiety (5.5±5.17) compared with the normative value (of 6.14±3.76), and higher for depression (4.15±4.0) compared with the normative value (of 3.68±3.07).
Arm/Group | HGG Patients
Number analyzed (Participants) | 10
Participants
  Leisure time I | 2
  Leisure time II | 2
  Leisure time III | 5
  Leisure time IV | 1

ADVERSE EVENTS:
Time Frame: adverse events were not monitored/assessed
Description: adverse events were not monitored/assessed
Arm/Group | HGG Patients
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2016-08-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT02965144/SAP_000.pdf
  • Informed Consent Form (2016-08-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT02965144/ICF_001.pdf
  • Study Protocol (2016-08-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT02965144/Prot_002.pdf